CLINICAL TRIAL: NCT03648983
Title: A Pilot Randomized Trial Comparing Arm Circumference and Bioimpedance Measurement for Early Detection and Treatment of Lymphedema in Patients Undergoing Axillary Lymph Node Dissection or Sentinel Node Biopsy
Brief Title: Arm Circumference Measurement With or Without Bioimpedance Spectroscopy in Finding Lymphedema Early in Patients With Stage I-III Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pi departure; service discontinued study
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-06-235; NCI-2014-01480 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-06-235E (Other: Albert Einstein College of Medicine); 11-047 (Other: Albert Einstein College of Medicine); LDEX (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2015-10-08; First posted 2018-08-28 (Actual); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-08

CONDITIONS: Lymphedema; Breast Cancer
Keywords: Enhanced Lymphedema
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard LE detection (Active Comparator): Arm measurements taken. Patients undergo arm circumference measurement at 4, 10, 16, 22, 28, and 34 months.
  Interventions: Procedure: arm circumference measurement
- Enhanced LE detection (Experimental): Bioimpedance spectroscopy used along with arm measurements. Patients undergo arm circumference measurement and bioimpedance spectroscopy at 4, 10, 16, 22, 28, and 34 months.
  Interventions: Procedure: arm circumference measurement; Device: Bioimpedance spectroscopy

INTERVENTIONS:
Procedure: arm circumference measurement — Undergo arm circumference measurement
Device: Bioimpedance spectroscopy — bioimpedance spectroscopy
  Other Names: BIS
  Arms: Enhanced LE detection

SUMMARY:
This randomized pilot clinical trial studies arm circumference measurement with or without bioimpedance spectroscopy in finding extra lymph node fluid build up in the arm (lymphedema) early in patients with stage I-III breast cancer undergoing lymph node dissection or sentinel node biopsy. Diagnostic procedures, such as bioimpedance spectroscopy, may allow doctors to find and diagnose lymphedema earlier than arm circumference measurement alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test, in a randomized controlled trial, the ability of the enhanced lymphedema (LE) detection program (ELED) versus arm circumference alone to detect early/reversible LE.

II. To compare the severity of LE in terms of changes in arm circumference at the site of greatest difference and L-Dex change, between the two detection modalities.

III. To assess the agreement between patients' self-report of swelling (mild, moderation and severe) and the extent of circumferential measurement/bioimpedance spectroscopy (BIS) difference.

IV. To compare the percentage of subjects with complete resolution of signs and symptoms of LE following treatment with a compression garment between the enhanced vs. standard detection groups.

V. To determine compliance with LE preventive care and treatment.

Patients are randomized to 1 of 2 arms: those undergo arm circumference measurement only and those undergoing undergo arm circumference measurement and bioimpedance spectroscopy. Measurements taken at 4, 10, 16, 22, 28, and 34 months.

In both arms, if lymphedema is diagnosed, patients are given a compression garment to wear daily for 6 weeks. If lymphedema does not improve after 6 weeks, patients undergo complete decongestive therapy over approximately 1 hour three times a week. Patients complete remedial exercises comprising active, repetitive range of motion of the involved extremity and light aerobic conditioning until extremity volume stabilizes or improves. Patients are also instructed to perform exercises at home.

After completion of study, patients diagnosed with lymphedema are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with stage I-III cancer of the female breast
* Patients scheduled to receive any type of radiation therapy to the breast or axilla are eligible; however, they must be registered to this study with pre-surgery measures taken prior to receiving neoadjuvant therapy as well as before surgery
* Patients scheduled to receive neoadjuvant chemotherapy are also eligible; however, they must be registered to this study with pre-surgery measurements taken prior to receiving neoadjuvant therapy as well as before surgery
* Patients with a history of other invasive malignancies are eligible as long as they have no evidence of disease 5 years post-diagnosis
* Patients with basal cell and squamous cell cancer of the skin are eligible
* Patients willing to return to the study site for the duration of the study (34 months)

Exclusion Criteria:

* Pregnant women
* Patients who are homebound or dependent upon a walker or wheelchair for mobility
* Patients diagnosed enhanced lymphedema
* Hypertensive patients who are using diuretics
* Documented cardiac conduction disturbances, unstable angina, dementia, or any other chronic disease which, in the opinion of the treating physician, significantly increases mortality over the next 2 years
* Prior history of carcinoma in situ, lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS), or invasive breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wiechmann, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.
Period: Overall Study
Arm/Group | Study Population
Started | 95
Completed | 0
Not Completed | 95
Not completed — Study was terminated due to PI departure | 95

BASELINE CHARACTERISTICS:
Population: Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.
Arm/Group | Study Population
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Enhanced Lymphedema Detection
Description: Rates of enhanced lymphedema detection will be compared between the enhanced versus standard detection groups with the Fisher's exact test. Adjustment for potential imbalances in patient characteristics will be accomplished by fitting logistic and Cox proportional hazards regression models.
  *** Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.***
Time Frame: During treatment (Up to 34 months)
Population: *** Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.***
Arm/Group | Study Population
Number analyzed (Participants) | 0

2. Secondary Outcome: Severity of Enhanced Lymphedema
Description: Severity of LE in terms of changes in arm circumference at the site of greatest difference and L-Dex change, will be compared between the enhanced versus standard detection groups with the Fisher's exact test. Adjustment for potential imbalances in patient characteristics will be accomplished by fitting logistic and Cox proportional hazards regression models.
Time Frame: During treatment (Up to 34 months)
Population: as for outcome 1
Groups:
- Study Population: *** Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.***
Arm/Group | Study Population
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Subjects With Complete Resolution of Signs of Enhanced Lymphedema
Description: The Fisher's exact test will be used to compare between the enhanced vs. standard detection groups the percentage of subjects with complete resolution of signs and symptoms of LE following treatment with a compression garment. Logistic regression models will also be fit to the data to adjust for potential confounders.
Time Frame: During treatment (up to 34 months) plus 1 year post treatment
Population: as for outcome 1
Arm/Group | Study Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: *** Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.***
Description: *** Study was terminated because PI left the institution. Study coordinator also left the institution. No data was analyzed. Participants' baseline records not available.***
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes